CLINICAL TRIAL: NCT03289468
Title: Study of Diagnosis of Color Power Doppler Combined Minimally Invasive Sampling for Endometrial Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2016T-14
Record Dates: First submitted 2017-06-15; First posted 2017-09-21 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-09

CONDITIONS: Endometrial Diseases
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — FirstXianJiaotongU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: Endometrial Benign Disease
  Interventions: Diagnostic Test: Voluson E8 (GE Medical Systems, USA), Minimally Invasive Endometrium Sampler
- Group2: Endometrial Cancer and Precancerous Lesions
  Interventions: Diagnostic Test: Voluson E8 (GE Medical Systems, USA), Minimally Invasive Endometrium Sampler

INTERVENTIONS:
Diagnostic Test: Voluson E8 (GE Medical Systems, USA), Minimally Invasive Endometrium Sampler — The endometrial thickness, basic characteristics information and endometrial blood flow energy index, endometrial vascularization index, blood flow index are detected by color power Doppler and the energy histogram of endometrium is obtained using a Voluson E8 (GE Medical Systems, USA) ultrasound system. The specimen of uterine cytology and endometrial tissue are obtained through minimally invasive endometrium sampler, which are diagnosed by pathology.

SUMMARY:
The postmenopausal women with vaginal bleeding were selected in this cross-sectional study. The basic characteristics information and endometrial blood flow energy index of endometrium were detected by color power Doppler ultrasound, and the energy histogram of endometrium was obtained. The specimen of uterine cytology and endometrial tissue were obtained through minimally invasive endometrium sampler, which were diagnosed by pathology. The statistical data were used to detect endometrial and precancerous lesions to observe the endpoint, and to provide the energy histogram model of the early warning endothelial diseases.

DETAILED DESCRIPTION:
The postmenopausal women with vaginal bleeding are selected in this cross-sectional study. The uterine bleeding in patients with blood system diseases, reproductive organ outside the uterus, other organs cancer metastasis to the uterus are excluded. The objects are divided into two groups(patients with endometrial benign diseases and patients with endometrial cancer and precancerous diseases) according to endometrial cytological and histological pathology. The endometrial thickness, basic characteristics information and endometrial blood flow energy index, endometrial vascularization index, blood flow index are detected by color power Doppler and the energy histogram of endometrium is obtained using a Voluson E8 (GE Medical Systems, USA) ultrasound system. Moreover,The specimen of uterine cytology and endometrial tissue are obtained through minimally invasive endometrium sampler, which were diagnosed by pathology.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with vaginal bleeding

Exclusion Criteria:

* Vaginal bleeding caused by hematological system diseases or genitals outside the uterus
* Uterine bleeding caused by other organ cancers metastasize to the uterus

Ages: 45 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with vaginal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The endometrial vascularization index | From March 2019 to December 2019
  The endometrial vascularization index include vascularization index(VI), flow index (FI) and vascularization flow index (VFI).

SECONDARY OUTCOMES:
The ultrasonography of endometrium | From March 2019 to December 2019
  The ultrasonography of endometrium included shape, boundary and echo.
The endometrial thickness | From March 2019 to December 2019
  The endometrial thickness in centimeter.
The blood flow index of endometrium | From March 2019 to December 2019
  The blood flow index include peak systolic velocity(PSV),cm/s, end diastolic velocity(EDV) ,cm/s, mean flow velocity(MnV) ,cm/s, pulsatility index(PI), resistance index(RI).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng YANG, Doctor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No